CLINICAL TRIAL: NCT01606293
Title: Use of Social Networking to Survey Women With Small and Large Cell Carcinomas of the Cervix
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0464
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Cervical Cancer
Keywords: Small cell carcinomas of the cervix; Large cell carcinomas of the cervix; Online surveys; Electronic surveys; Questionnaires; Facebook; Social networking support groups
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carcinomas of the Cervix Survey: Women with small and large cell carcinomas of the cervix, who are members of the Facebook group found at the uniform resource locator https://www.facebook.com/SmallCellCC through an online link.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Completion of online surveys taking approximately 15 - 20 minutes.
  Other Names: Electronic surveys

SUMMARY:
Objectives:

Primary: 1. To assess the feasibility of using social networking groups to survey patients with rare cancers.

Secondary:1. To elucidate the current means for diagnosis and treatment of women with small and large cell carcinomas of the cervix. 2. To evaluate anxiety regarding diagnosis, treatment, and recurrence among women with small and large cell carcinomas of the cervix.

DETAILED DESCRIPTION:
The entire study will be conducted electronically. A survey assessing presentation of disease, treatment history and follow-up (appendix A) will be hosted on a secured online server. In addition respondents will be asked to complete a battery of 40 questions assessing anxiety regarding their diagnosis and fear of recurrence based on previously published instruments (appendix B).

Patients will be asked to provide data on the presenting symptoms at the time of the diagnosis, method of diagnosis, HPV detection, modalities used as initial treatment, specialty of the physician administering the treatment, stage, follow up interval and diagnostic studies, recurrence free interval and treatments offered/received at the time of recurrence.

To assess anxiety and fear of recurrence we will be using questions from instruments initially used in a breast cancer population:

The Concerns About Recurrence Scale (CARS): The CARS has two main parts. In the first part, overall fear of recurrence is assessed with four questions addressing frequency, potential for upset, consistency, and intensity of fears. Participants rate each of these items on a 1-to-6 scale. In the second part, the nature of women's fears about recurrence is assessed with 26 items that follow the stem phrase: "I worry that a recurrence of cancer would" Participants use a 5-pointscale, ranging from 0 (not at all), to 1 (a little), to 2 (moderately), to 3 (a lot), and to 4 (extremely), to indicate the extent to which they worry about each item.

Lerman Cancer Worry Scale: This includes three items, one measuring the frequency of worrying about "getting recurrence cancer someday," and two items measuring the impact of worry on mood and performing daily activities. For cancer worry, subjects will rate their current levels of worry about getting cancer recurrence someday on a 5-point scale with points labeled not at all (1), rarely (2), sometimes (3), often (4), and almost all the time (5). For impact of worry on mood and on functioning, respondents experiencing cancer worries will rate the current impact of such worries on their moods and on their ability to perform their daily activities using a 4-point scale with points labeled not at all (I),a little (2), somewhat (3), and a lot (4).

The Survey will be offered to all patients who are members of the Facebook group found at the uniform resource locator https://www.facebook.com/SmallCellCC through an online link. We expect the survey to take participants 15-20 minutes to complete. Surveys with similar anxiety measuring elements conducted by phone and on the internet have been reported with success.

Patients will be presented with an online informed consent prior to taking the survey. In addition patients will be provided with an email address and a phone number to use if they have any questions or wish to withdraw from the study. Upon reading the informed consent patients will be able to proceed to the questionnaire hence signifying their informed consent or back to Facebook indicating their refusal. No personal identifying data will be collected. Prior to taking the survey they will be given a serial number to associate with their answers in case they wish to withdraw in the future.

ELIGIBILITY:
Inclusion Criteria:

* Women with small cell carcinoma of the cervix who are members of a social networking support group on Facebook who give informed consent and are able to complete a 15 min online survey.

Exclusion Criteria:

* Women with small cell carcinoma of the cervix who are members of a social networking support group on Facebook who cannot respond to an English online survey.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are members of the Facebook group found at the uniform resource locator https://www.facebook.com/SmallCellCC through an online link.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05-24 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Using Social Networking Groups to Survey Patients with Rare Cancers. | 1 day
  The entire study will be conducted electronically. A survey assessing presentation of disease, treatment history and follow-up will be hosted on a secured online server. In addition respondents will be asked to complete a battery of 40 questions assessing anxiety regarding their diagnosis and fear of recurrence based on previously published instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Frumovitz, MD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org